CLINICAL TRIAL: NCT03582566
Title: Training-Induced Language and Literacy Improvement in Children With Cochlear Implants
Brief Title: Training Language and Literacy for Children Who Use CIs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Northwestern University (Other)
Responsible Party: Principal Investigator, erin ingvalson, Associate Professor, Florida State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 037312
Record Dates: First submitted 2018-06-18; First posted 2018-07-11 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Hearing Loss, Sensorineural
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Intervention Model Description: The efficacy of phonological awareness (Earobics) and working memory (Cogmed) training alone and in combination are compared to an active control (Splashmath).
Who Masked: Outcomes Assessor
Masking Description: Assessors are blind to treatment condition. Intervention providers are blind to assessment outcomes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phonological Awareness (Experimental): Children will play games to practice their rhyming, sound sequencing, and letter-sound knowledge. These games are all implemented in the Earobics program.
  Interventions: Behavioral: Phonological Awareness
- Working Memory (Experimental): Children will play games designed to help them hold and manipulate objects in memory. These games are implemented in Cogmed.
  Interventions: Behavioral: Working Memory
- Phonological Awareness + Working Memory (Experimental): Children will practice both their sound skills (Earobics) and their memory skills (Cogmed).
  Interventions: Behavioral: Phonological Awareness + Working Memory
- Active Control (Active Comparator): Children will play games to practice their addition and subtraction skills (Splashmath).
  Interventions: Behavioral: Active Control

INTERVENTIONS:
Behavioral: Phonological Awareness — Earobics training
  Arms: Phonological Awareness
Behavioral: Working Memory — Cogmed training
  Arms: Working Memory
Behavioral: Phonological Awareness + Working Memory — Earobics + Cogmed training
  Arms: Phonological Awareness + Working Memory
Behavioral: Active Control — Spashmath
  Arms: Active Control

SUMMARY:
This study aims to determine the effectiveness of computer games to improve language and literacy outcomes for children who have hearing loss. Children will be assigned to one of four conditions: phonological awareness training, working memory training, phonological awareness + working memory training, or active control.

DETAILED DESCRIPTION:
Both phonological awareness and working memory are known to be important for children's language and literacy learning. Though there are computer games that claim to improve phonological awareness and working memory, it is unknown if these games will improve language and literacy skills for children who have hearing loss.

The investigators will first determine if the games are effective for improving language and phonological awareness in children with hearing loss relative to an active control condition. Secondly, the investigators will determine if gains in phonological awareness and working memory translate into gains in language and literacy skills relative to active control.

ELIGIBILITY:
Inclusion Criteria:

* Prelingual hearing loss
* Use of amplification device (hearing aid and/or cochlear implant) for at least one year
* Able to visit the clinic 3x/week for 12 weeks

Exclusion Criteria:

* No developmental delays (Down's syndrome, Autism spectrum disorder)

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2023-06 (Actual); Study Completion 2023-06 (Actual)

PRIMARY OUTCOMES:
Change in Phonological Awareness Test scores | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of phonological awareness. Scores are from 0-100 with higher scores indicating better performance.
Change inComprehensive Test of Phonological Awareness | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of phonological awareness. Scores are from 0-100 with higher scores indicating better performance.
Change in Children's Test of Nonword Repetition | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of verbal working memory

SECONDARY OUTCOMES:
Change in Oral Written Language Scales | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of language and literacy skills. Measures performance on expressive and receptive language, and reading and writing abilities. Scores are age-adjusted.
Change in Receptive/Expressive One Word Picture Vocabulary Test | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of vocabulary knowledge. Scores are from 0-100 with higher scores indicating better performance.
Change in Woodcock Johnson Reading Mastery Test | Baseline, post-intervention (8 weeks post-baseline), 6 months post-baseline
  Change in a standardized test of early literacy skills. Scores are from 0-100 with higher scores indicating better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Ingvalson, PhD, Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Northwestern University, Evanston, Illinois